CLINICAL TRIAL: NCT06607757
Title: Phase II Neoadjuvant Study Evaluating Capivasertib Plus Fulvestrant vs Fulvestrant in Patients With Primary High-risk Lobular Breast Cancer- LOBSTER
Brief Title: Capivasertib Plus Fulvestrant vs. Fulvestrant in Primary High-risk Lobular Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBG118 - LOBSTER; 2023-509292-17-00 (EU CTIS Number)
Record Dates: First submitted 2024-06-14; First posted 2024-09-23 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: CCCA Assessed by Ki67 Drop Below <2.7% From Baseline
MeSH Terms: interventions — capivasertib; Fulvestrant

STUDY DESIGN:
Intervention Model Description: Evaluation of treatment outcome
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Capivasertib (400 mg po twice daily d1-4 followed by 3 days off) for 2 weeks followed by capivasertib (400 mg po twice daily d1-4 followed by 3 days off) and fulvestrant (500 mg i.m. q28d, with an additional 500 mg dose given two weeks after the initial dose) for additional 8 weeks (overall 4 administrations of fulvestrant)
  Interventions: Drug: Capivasertib; Drug: Fulvestrant injection
- Arm B (Active Comparator): Fulvestrant (500mg i.m. q28d, with an additional 500 mg dose given two weeks after the core biopsy and the initial dose) for 10 weeks (overall 4 administrations)
  Interventions: Drug: Fulvestrant injection

INTERVENTIONS:
Drug: Capivasertib — find arm A description
  Other Names: Truqap
  Arms: Arm A
Drug: Fulvestrant injection — find arm B description
  Other Names: Faslodex

SUMMARY:
This is a multicenter, prospective, open-label, randomized phase II study to evaluate the CCCA assessed by Ki67 drop below <2.7% from baseline to week 2 (window of opportunity) and to week 10 with capivasertib plus fulvestrant compared with fulvestrant alone as neoadjuvant treatment for primary high-risk lobular breast cancer patients.

120 patients will be randomized to receive:

- Capivasertib (400 mg po twice daily d1-4 followed by 3 days off) for 2 weeks followed by capivasertib (400 mg po twice daily d1-4 followed by 3 days off) and fulvestrant (500 mg i.m. q28d, with an additional 500 mg dose given two weeks after the initial dose) for additional 8 weeks (overall 4 administrations of fulvestrant)

or

- Fulvestrant (500mg i.m. q28d, with an additional 500 mg dose given two weeks after the core biopsy and the initial dose) for 10 weeks (overall 4 administrations) Treatment will be given until surgery/core-biopsy, disease progression, unacceptable toxicity, or withdrawal of consent of the patient.

All patients will undergo core-biopsies, under treatment and after completing study therapy in order to assess Ki67%. Further treatment including surgery, (neo)adjuvant chemotherapy, radiotherapy, and (neo)adjuvant endocrine therapy will be administered at the discretion of the investigator and according to standard of care outside the clinical trial.

DETAILED DESCRIPTION:
The evaluation of CCCA in the HR+/HER2- invasive lobular breast cancer patient population allows assessment of treatment efficacy with an achievable sample size of HR+/HER2- breast cancer patients within an acceptable and scientifically meaningful duration of recruitment. CCCA can be assessed immediately after last patients end of treatment. Central blinded pathological assessment of CCCA is planned in this study as a standardized preparation of the sampled tissue by the central pathologist. This pathologist is blinded regarding the study therapy administered, i. e. with or without capivasertib.

The addition of capivasertib to fulvestrant in many clinical trials correlates with an improvement in PFS compared to fulvestrant alone in patients with HR+/HER2- locally advanced or metastatic breast cancer. This effect was observed regardless of a PI3K/AKT/mTOR pathway activation. None of the ongoing studies investigate the effects of the combined treatment in invasive lobular breast cancer. Given that these tumors are less likely to respond to chemotherapy, identification of patients that can be spared from chemotherapy is desirable. On the other hand, it is important to identify patients with invasive lobular breast cancer not responding to neoadjuvant ET who might be at increased risk for recurrence, who would therefore potentially benefit from further adjuvant therapies including chemotherapy.

Given the high rates of PI3K pathway alterations in such tumors, it is expected that the CCCA rate could be increased by adding capivasertib to fulvestrant. GBG expect that the potential benefit of improved CCCA rate with a combination treatment compared to fulvestrant monotherapy would outweigh the potential risks due to added toxicity, which has already been shown in clinical trials to be well tolerated by patients.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to beginning specific protocol procedures, including expected cooperation of the patients for the treatment and followup, and documented according to the local regulatory requirements.
2. Postmenopausal women with age at diagnosis ≥ 18 years.

   Postmenopausal status is defined as:
   * Age ≥60 years
   * Age <60 years and amenorrhea for at least 12 continuous months with no identified cause other than menopause
   * Bilateral oophorectomy Negative pregnancy test (urine or serum) within 14 days prior to randomization for all postmenopausal women 50 years of age or younger without bilateral oophorectomy
3. Unilateral or bilateral primary untreated lobular invasive carcinoma of the breast. In case of bilateral breast cancer, both sides must be lobular; the lead tumor has to be defined by the investigator based on the inclusion criteria for the respective subtype and the risk status. Lobular histology has to be centrally confirmed.
4. Willingness and ability to provide archived formalin fixed paraffin embedded (FFPE) tissue block from core biopsy before the start of neoadjuvant therapy.
5. Centrally confirmed HER2-negative (IHC score 0-1+ or ISH negative according to ASCO/CAP guideline) and HR-positive (≥10% positive stained cells) disease, assessed on the core of diagnostic biopsy. Ki67% >10% is required. In case of bilateral breast cancer, HER2-negative, HR-positive and lobular histology status has to be confirmed for both sides.
6. Patients with invasive lobular breast cancer at high risk for recurrence defined as cT1c and clinical nodal involvement (cN+) or ≥ cT2 disease (irrespective of nodal involvement).
7. No clinical evidence of distant metastases.
8. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.
9. Estimated life expectancy of at least 5 years irrespective of the diagnosis of breast cancer.
10. The patient must be accessible for scheduled visits, treatment, and followup.
11. Normal cardiac function must be confirmed according to local guidelines.
12. Laboratory requirements:

    Hematology
    * Absolute neutrophil count (ANC) ≥1.5 x 109 / L
    * Platelets ≥100 x 109 / L
    * Hemoglobin ≥10 g/dL (≥6.2 mmol/L) Hepatic function
    * Total bilirubin <1.25x ULN
    * AST and ALT <=1.5x ULN
    * Alkaline phosphatase <=2.5x ULN Glucose Metabolism
    * HbA1c <8.0% (63.9 mmol/mol) Renal Function
    * Creatinine <1.25x ULN or creatinine clearance ≥50 ml/min (if creatinine is above ULN according to Cockroft-Gault)
13. Complete staging work-up prior to the initiation of neoadjuvant therapy as per standard recommendations.

Exclusion Criteria:

1. Female patients of childbearing potential.
2. Excisional biopsy or lumpectomy performed prior to study entry.
3. Surgical axillary staging procedure including sentinel lymph node biopsy prior to randomization. Exceptions: FNA or core biopsy of an axillary lymph node.
4. Any previous treatment including endocrine therapy, chemotherapy, radiotherapy or targeted therapy (including AKT inhibitor or PIK3 inhibitor) for the currently diagnosed breast cancer.
5. Concurrent use of herbal or natural products intended as treatment or prophylaxis for any type of cancer.
6. Known hypersensitivity reaction to one of the compounds or substances used in this protocol.
7. Potent inhibitors or inducers of CYP3A4 within 2 weeks prior to the first dose of study treatment (3 weeks for St John's wort).
8. Refractory nausea and vomiting, chronic gastrointestinal disease, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption, distribution, metabolism, or excretion of capivasertib.
9. Any contraindication for fulvestrant.
10. Patients with definitive clinical or radiologic evidence of stage IV cancer (metastatic disease) are not eligible.
11. Patients with a history of any malignancy are ineligible with the following exceptions:

    * Patient has been disease-free for at least 5 years and is at low risk for recurrence of that malignancy except for breast cancer.
    * CIS of the cervix, basal cell and squamous cell carcinomas of the skin.
12. History of type I or type II diabetes mellitus requiring insulin.
13. Severe and relevant co-morbidity that would interact with the application of study drugs or the participation in the study, including cerebrovascular incident including transient ischemic attack, or symptomatic pulmonary embolism, active infection requiring intravenous anti-microbial treatment (antibiotics, anti-fungal, and anti-viral drugs) within 1 week of enrolment. Patients with confirmed Gilbert's syndrome may be included in the study.
14. Known medically history of HIV infection, tuberculosis, or hepatitis B.
15. History of and/or active cardiac disease that would preclude the use of study treatments. This includes but is not confined to any of the following cardiac criteria:

    * Clinically significant cardiac dysfunction including heart failure (NYHA II-IV), active ventricular arrhythmias requiring medication or arrhythmias requiring a pacemaker, and history of a myocardial infarction within 6 months prior to randomization, angina pectoris, atrial fibrillation of any grade, coronary/peripheral artery bypass graft, angioplasty, or vascular stent.
    * Mean resting QT interval corrected by Fridericia's formula (QTcF) >470 msec obtained from 3 consecutive ECGs.
    * Increased risk of QTc prolongation or risk of arrhythmic events such as heart failure, uncontrolled electrolyte disorders (e.g., hypocalcemia, hypokalemia, or hypomagnesemia), potential for torsades de pointes, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age, or any concomitant medication known to prolong the QT interval.
16. Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving therapy.
17. History of significant neurological or psychiatric disorders including psychotic disorders, dementia, or seizures that would prohibit the understanding and giving of informed consent.
18. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results (such as severe or uncontrolled systemic diseases, including uncontrolled hypertension or hypotension (BP <50mmHg), significant aneurysm, renal transplant and active bleeding diseases).
19. Major surgical procedure (excluding placement of vascular access) or significant traumatic injury within 4 weeks of the first dose of study intervention or an anticipated need for major surgery during the study.
20. Participation in another clinical study with a study intervention or investigational medicinal device administered in the 4 weeks prior to first dose of study intervention or concurrent enrolment in another clinical study unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
To assess complete cell cycle arrest (CCCA). | Up to 14 weeks
  The primary endpoint CCCA is defined as Ki67 drop to <2.7% after approximately 10 weeks (will be assessed centrally on the breast tissue submitted to central pathology)

SECONDARY OUTCOMES:
To asses safety and tolerability | Up to 14 weeks
  Tolerability and safety analyses include assessment of patients whose treatment had to be dose reduced, delayed or permanently stopped.
To assess patholgogical complete response rate (pCR) by different definitions | Up to 14 weeks
  Pathological complete response (pCR ypT0 ypN0) is defined as no microscopic evidence of residual invasive and non-invasive viable tumor cells in all resected specimens of the breast and axilla.
To assess breast conservation rate (BCS) | Up to 14 weeks
  BCS is defiened as tumorectomy, segmentectomy or quandrantectomy as the most radical surgery.
To assess invasive disease-free survival (iDFS) and overall survival (OS) | through study completion, an average of 2 years
  iDFS is defined as time from randomization until first iDFS event OS is defined as time from randomization until death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Sibylle Loibl, Prof. Dr. med., Principal Investigator — ESMO, ASCO, AGO Kommission Mamma (member); Goethe University Frankfurt; GBG Forschungs GmbH
Locations (25):
- Germany (25):
  - Haematologie-Onkologie im Zentrum MVZ GmbH, Augsburg
  - Charité, Berlin
  - Onkologische Schwerpunktpraxis - Studiengesellschaft Onkologie Bielefeld GbR, Bielefeld
  - Hämato-Onkologie im Medicum - Onkologie und Hämatologie, Bremen
  - Kliniken der Stadt Köln GmbH - Brustzentrum Köln-Holweide, Cologne
  - Carl-Thiem-Klinikum gGmbH - Frauenklinik, Cottbus
  - Kath. St. Paulus GmbH - Klinische Forschung, Dortmund
  - Universitätsklinikum Essen - Klinik für Frauenheilkunde und Geburtshilfe, Essen
  - Klinikum Frankfurt Höchst GmbH - Klinik für Gynäkologie und Geburtshilfe, Frankfurt am Main
  - Praxis für Interdisziplinäre Onkologie & Hämatologie, Freiburg im Breisgau
  - Mammazentrum Hamburg - am Krankenhaus Jerusalem, Hamburg
  - Universitätsklinikum des Saarlandes - Frauenklinik, Homburg
  - Klinikum Kassel GmbH - Frauenklinik, Kassel
  - St. Elisabethen-Krankenhaus gGmbH - Senologie / Brustzentrum, Leipzig
  - Medizinisches Versorgungszentrum MediaVita GmbH Muenster, Münster
  - Klinikum Oldenburg AöR - Universitätsklinik für Innere Medizin - Onkologie, Oldenburg
  - MVZ für Hämatolgie und Onkologie Ravensburg GmbH - Studienzentrum, Ravensburg
  - Klinikum Südstadt - Universitätsfrauenklinik, Rostock
  - Leopoldina-Krankenhaus der Stadt Schweinfurt - Frauenklinik, Schweinfurt
  - Johanniter-Krankenhaus Genthin-Stendal - Klinik für Frauenheilkunde und Geburtshilfe, Stendal
  - Kreiskrankenhaus Torgau - Gynäkologie, Torgau
  - Praxisnetzwerk Haematologie und internistische Onkologie Ueberoertliche Berufsausuebungsgemeinschaft - Hämatologie und Onkologie, Troisdorf
  - Marienhospital Witten - Brustzentrum, Witten
  - Klinikum Worms gGmbH - Frauenklinik, Worms
  - Helios Klinikum Wuppertal GmbH - Landesfrauenklinik, Wuppertal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rugo HS, Oliveira M, Howell SJ, Dalenc F, Cortes J, Gomez HL, Hu X, Jhaveri KL, Krivorotko P, Loibl S, Morales Murillo S, Nowecki Z, Okera M, Park YH, Sohn J, Toi M, Iwata H, Yousef S, Zhukova L, Logan J, Twomey K, Khatun M, D'Cruz CM, Turner NC. Capivasertib and fulvestrant for patients with hormone receptor-positive advanced breast cancer: characterization, time course, and management of frequent adverse events from the phase III CAPItello-291 study. ESMO Open. 2024 Sep;9(9):103697. doi: 10.1016/j.esmoop.2024.103697. Epub 2024 Sep 5. PMID 39241495
- See also: GBG Website with information about LOBSTER Trial — https://www.gbg.de/studien/lobster